CLINICAL TRIAL: NCT01540630
Title: A Phase IIa Placebo-Controlled, Double-Blind Randomized Withdrawal Study to Evaluate the Safety and Efficacy of CNV1014802 in Patients With Trigeminal Neuralgia
Brief Title: A Phase IIa Withdrawal Study of CNV1014802 in Patients With Trigeminal Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNV1014802/202
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — vixotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CNV1014802 (Experimental)
  Interventions: Drug: CNV1014802
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNV1014802 — CNV1014802 150mg tid for 28 days. Dose may be increased to 350mg bid following interim evaluation of efficacy.
  Arms: CNV1014802
Drug: Placebo — Double-blind placebo comparator for 28 days.
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized withdrawal study comparing CNV1014802 with placebo in patients with trigeminal neuralgia who have successfully responded to CNV1014802 in an initial open-label phase.

Patients will participate in an initial open-label treatment period of 21 days of CNV1014802 150mg three times a day (tid). Responders will be randomized to 28 days of CNV1014802 150mg tid or placebo.

Following an interim analysis after 10 evaluable patients have completed the open-label phase, the dose regimen may be increased to 350mg twice a day (bid) for the remainder of the trial if the responder rate is less than 60%.

DETAILED DESCRIPTION:
In order to be randomised and enter the double-blind placebo controlled phase of the study, patients must satisfy at least one of the following criteria:

* 30% or more decrease in number of paroxysms (either spontaneous, evoked, or both)
* 30% reduction in the severity of pain experienced during the paroxysm (either spontaneous, evoked or both)
* A Patient Global Improvement of Change rating of much improved/very much improved The response will be compared with the baseline recordings of pain made in the 7 day run-in period. If a patient meets one of these criteria they are termed a responder, and will be eligible to be randomized into the double-blind treatment phase.

During the double-blind randomised phase, patients will be evaluated to determine if they meet the failure criteria at each clinic visit which will occur every 7 days in the double-blind treatment period. The number of failures on CNV1014802 versus number of failures on placebo during the double-blind treatment period will be the primary outcome of the study.

Patients will be classified as a treatment failure if they meet one of the following criteria:

* 50% increase in the frequency of paroxysms compared to the final 7 days of the open-label period
* 50% increase in the severity of pain experienced in the paroxysms compared to the final 7 days of the open-label period
* A Patient Global Improvement of Change rating of much worse/very much worse
* The patient discontinues the study due to 'Lack of Efficacy'
* The patient discontinues due to an adverse reaction or poor tolerability considered to be related to study medication

This study was previously posted by Convergence Pharmaceuticals, Ltd., which has been acquired by Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 70 years, with a diagnosis of trigeminal neuralgia; IHS criteria to be used.
* Female patients must be of non-child bearing potential or agree to use an approved form of contraception
* Male patients must agree to use an approved form of contraception
* Body weight > 50 kg for men and > 45 kg for women.
* BMI ≤ 34.9
* Capable of giving written informed consent. Informed consent must be obtained prior to the commencement of any study related procedures.
* QTcB either/or QTcF < 450 msec in two of three ECGs conducted at screening
* AST and ALT < 2xULN; alkaline phosphatase and bilirubin < 1.5xULN.
* Approved concomitant medications must have been stable for at least 3 weeks prior to day 0.

Exclusion Criteria:

* Patients who are known non-responders to sodium channel blockers at therapeutic doses.
* Patients with causes for their facial pain other than that specified in Inclusion Criterion
* A positive pre-study drug screen.
* A positive history of HIV.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* History of any liver disease within the last 6 months, with the exception of known Gilbert's disease.
* History of excessive regular alcohol consumption within 6 months of the study.
* Patients with a history or risk of seizures or a history of epilepsy, head injury or related neurological disorders
* Patients with a history of uncontrolled or poorly controlled hypertension, with systolic BP frequently exceeding 160mmHg and/or diastolic BP frequently exceeding 100mmHg, or patients who have BP greater than or equal to 160mmHg systolic and/or greater than or equal to 100mmHg diastolic at screening after repeated measurements
* History or presence of significant cardiovascular, gastro-intestinal, or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Patients with conditions known to affect cardiac conduction or a personal or familial history of Brugada syndrome
* Pregnant females or lactating females.
* History or presence of any clinically significant abnormality in vital signs/ECG/laboratory tests or have any medical or psychiatric condition, which, in the opinion of the Investigator may interfere with the study procedures or compromise patient safety.
* History of suicidal ideation and/or suicide attempts or clinical evidence of recent major depression.
* Patients who are unable to maintain approved medications for their trigeminal neuralgia at a stable dose during the study.
* Unable to refrain from excessive use of sedatives.
* Unable to comply with the prohibited concomitant medication restrictions as detailed in the protocol. This includes but is not limited to sodium channel blockers or drugs that adversely interact with a monoamine oxidase-B inhibitor: MAOI's, antidepressants, opioids and sympathomimetic agents.
* History of hypersensitivity to CNV1014802.
* The patient has participated in a clinical trial and has received an investigational product within 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) prior to the start of this study.
* Exposure to more than four new chemical entities (medications for which no marketing authorization has been obtained) within 12 months prior to the first dosing day.
* Where participation in the study would result in total donation of blood or blood products in excess of 500mL within a 56 day period.
* Patient is mentally or legally incapacitated.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-03-31 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
The number of failures on CNV1014802 vs. number of failures on placebo during the double-blind treatment period will be the primary outcome of the study. | 4 weeks
  Patients will be classified as a treatment failure if they meet one of the following criteria:
  * 50% increase in the frequency of paroxysms compared to the final 7 days of the open-label period
  * 50% increase in the severity of pain experienced in the paroxysms compared to the final 7 days of the open-label period
  * A Patient Global Improvement of Change rating of much worse/very much worse
  * The patient discontinues the study due to 'Lack of Efficacy'. v. The patient discontinues due to an adverse reaction or poor tolerability considered to be related to study medication

SECONDARY OUTCOMES:
Secondary pain endpoints | 4 weeks
  * Number and severity of paroxysms of pain in the 21 day open-label period, both evoked and spontaneous
  * Average 24 hour pain intensity numerical rating scale (PI-NRS)
  * Patient and Physician Clinical Global Impression of Change
  * Brief Pain Inventory - Facial

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Professor Joanna Zakrzewska, London, United Kingdom

REFERENCES:
- [Background] Zakrzewska JM, Palmer J, Ettlin DA, Obermann M, Giblin GM, Morisset V, Tate S, Gunn K. Novel design for a phase IIa placebo-controlled, double-blind randomized withdrawal study to evaluate the safety and efficacy of CNV1014802 in patients with trigeminal neuralgia. Trials. 2013 Nov 23;14:402. doi: 10.1186/1745-6215-14-402. PMID 24267010
- [Derived] Zakrzewska JM, Palmer J, Bendtsen L, Di Stefano G, Ettlin DA, Maarbjerg S, Obermann M, Morisset V, Steiner D, Tate S, Cruccu G. Challenges recruiting to a proof-of-concept pharmaceutical trial for a rare disease: the trigeminal neuralgia experience. Trials. 2018 Dec 27;19(1):704. doi: 10.1186/s13063-018-3045-1. PMID 30587219
- [Derived] Zakrzewska JM, Palmer J, Morisset V, Giblin GM, Obermann M, Ettlin DA, Cruccu G, Bendtsen L, Estacion M, Derjean D, Waxman SG, Layton G, Gunn K, Tate S; study investigators. Safety and efficacy of a Nav1.7 selective sodium channel blocker in patients with trigeminal neuralgia: a double-blind, placebo-controlled, randomised withdrawal phase 2a trial. Lancet Neurol. 2017 Apr;16(4):291-300. doi: 10.1016/S1474-4422(17)30005-4. Epub 2017 Feb 17. PMID 28216232
- See also: EudraCT Tabulated Result — https://www.clinicaltrialsregister.eu/ctr-search/trial/2010-023963-16/results